CLINICAL TRIAL: NCT05209997
Title: An Observational, Multicenter, National Study with Real-life Retrospective Data Collection on the Combined Use of Sibutramine and Topiramate As Anti-obesity Treatment in Overweight Patients with Comorbidity(ies) or Obesity.
Brief Title: Observational, Real-life, Retrospective, Data Collection, Use Sibutramine/topiramate in Overweight Comorbidities/obesity
Acronym: TOLERASIT
Status: Withdrawn | Type: Observational
Why Stopped: The study was withdrawn following a thorough evaluation of the current scientific landscape and ongoing advancements in the field. This decision was made to ensure that the research remains aligned with the highest standards of innova
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: EF179
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Source document data collection — Data from all adult patients, of both sexes, for whom combination treatment with sibutramine and topiramate, both at any dose/dosage, were prescribed between the year 2011 and the beginning of the study will be colected in the study.

SUMMARY:
An observational, multicenter, national study with retrospective real-life data collection on the combined treatment of sibutramine and topiramate (off-label use) for the treatment of overweight with comorbidity(ies) or obesity. Data from all adult patients, of both sexes, for whom combination treatment with sibutramine and topiramate, both at any dose/dosage, were prescribed between the year 2011 and the beginning of the study will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Both sexes
* Diagnose of overweight with comorbidity(ies) or obesity
* Treatment use of sibutramine combined with topiramate
* Treatment prescription between 2011 and the beginning of the study

Exclusion Criteria:

* Use of topiramate for other condition besides overweight with comorbidity(ies) or obesity
* Individual use of one of the medications (sibutramine or topiramate)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, of both sexes, for whom combination treatment with sibutramine and topiramate, both at any dose/dosage, with prescribed treatment between the year 2011 and the beginning of the study
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients who achieved a weight loss greater than 5% | 20 years
  Identification of the percentage of patients who achieved a weight loss greater than 5% in relation to the initial body weight.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Eurofarma Laboratórios S.A, São Paulo, São Paulo
  - HC-FMUSP, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No